CLINICAL TRIAL: NCT01186991
Title: A Randomized, Phase II, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Onartuzumab And/or Bevacizumab in Combination With Paclitaxel in Patients With Metastatic, Triple-Negative Breast Cancer
Brief Title: Study Evaluating the Safety and Efficacy of Onartuzumab And/or Bevacizumab in Combination With Paclitaxel in Participants With Metastatic, Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OAM4861g; GO01334 (Other: Hoffmann-La Roche); 2010-020101-32 (EudraCT Number)
Record Dates: First submitted 2010-08-09; First posted 2010-08-23 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — onartuzumab; Bevacizumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Onartuzumab + Bevacizumab + Paclitaxel (Experimental): Participants will receive treatment with onartuzumab, bevacizumab, and paclitaxel, which may continue until disease progression, unacceptable drug-related toxicity, investigator decision, death, or completion of study, whichever occurs first (up to approximately 5 years).
  Interventions: Drug: Onartuzumab; Drug: Bevacizumab; Drug: Paclitaxel
- Onartuzumab + Placebo + Paclitaxel (Experimental): Participants will receive treatment with onartuzumab, placebo matching to bevacizumab, and paclitaxel, which may continue until disease progression, unacceptable toxicity, investigator decision, death, or completion of study, whichever occurs first (up to approximately 5 years).
  Interventions: Drug: Onartuzumab; Drug: Paclitaxel; Drug: Bevacizumab Placebo
- Placebo + Bevacizumab + Paclitaxel (Active Comparator): Participants will receive treatment with placebo matching to onartuzumab, bevacizumab, and paclitaxel, which may continue until disease progression, unacceptable toxicity, investigator decision, death, or completion of study, whichever occurs first (up to approximately 5 years).
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Onartuzumab Placebo

INTERVENTIONS:
Drug: Onartuzumab — Onartuzumab will be administered as intravenous (IV) infusion at a dose of 10 milligrams per kilogram (mg/kg) on Day 1 and Day 15 of each 28-day cycle. The dose of onartuzumab will be based on the participant's weight at screening and will remain the same throughout the study.
  Other Names: MetMAb
  Arms: Onartuzumab + Bevacizumab + Paclitaxel; Onartuzumab + Placebo + Paclitaxel
Drug: Bevacizumab — Bevacizumab will be administered as IV infusion at a dose of 10 mg/kg on Day 1 and Day 15 of each 28-day cycle. The dose of bevacizumab will be based on the participant's weight at screening and will remain the same throughout the study.
  Other Names: Avastin
  Arms: Onartuzumab + Bevacizumab + Paclitaxel; Placebo + Bevacizumab + Paclitaxel
Drug: Paclitaxel — Paclitaxel will be administered as IV infusion at a dose of 90 milligrams per meter-squared (mg/m^2) on Day 1, Day 8, and Day 15 of each 28-day cycle.
  Other Names: Taxol
Drug: Bevacizumab Placebo — Placebo matching to bevacizumab will be administered as IV infusion on Day 1 and Day 15 of each 28-day cycle.
  Arms: Onartuzumab + Placebo + Paclitaxel
Drug: Onartuzumab Placebo — Placebo matching to onartuzumab will be administered as IV infusion on Day 1 and Day 15 of each 28-day cycle.
  Arms: Placebo + Bevacizumab + Paclitaxel

SUMMARY:
This is a randomized, Phase II, double-blind, multicenter, placebo-controlled trial designed to preliminarily estimate the efficacy and evaluate the safety and tolerability of onartuzumab (MetMAb) + bevacizumab + paclitaxel and onartuzumab + placebo + paclitaxel versus placebo + bevacizumab + paclitaxel in participants with metastatic or locally recurrent, triple-negative breast cancer who either have not received treatment (first-line) or have progressed after one conventional cytotoxic chemotherapy regimen (second-line).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Histologically confirmed estrogen receptor (ER)-, progesterone receptor (PR)-, and human epidermal growth factor 2 (HER2)-negative (triple-negative) adenocarcinoma of the breast
* Confirmed availability of tumor tissue

Exclusion Criteria:

* Prior therapy with two or more regimens for metastatic breast cancer
* Any systemic anti-cancer therapy within 3 weeks prior to Day 1 of Cycle 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 30 days prior to Day 1 of Cycle 1
* Prior therapy with a taxane for metastatic breast cancer
* Prior therapy with bevacizumab, sorafenib, sunitinib, or other putative vascular endothelial growth factor (VEGF) pathway-targeted therapy following diagnosis of breast cancer
* Prior therapy with hormones and/or trastuzumab
* Inadequate hematology, renal, or hepatic organ function

Bevacizumab Exclusion Criteria:

* Uncontrolled hypertension (systolic pressure greater than [>] 150 millimeters of mercury [mmHg] and/or diastolic pressure > 100 mmHg), with or without anti-hypertensive medication
* Evidence of bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Participants Who Have not Received Prior Systemic Therapy or Have Progressed to Prior First-line Treatment | From randomization until disease progression (PD), relapse, or death on study (within 30 days of last study drug administration) from any cause, whichever occurs first (to be assessed according to local standard of care overall up to 5 years)

SECONDARY OUTCOMES:
PFS According to RECIST v1.1 in Participants Who Have not Received Prior Systemic Therapy | From randomization until PD, relapse, or death on study from any cause, whichever occurs first (to be assessed according to local standard of care overall up to 5 years)
Percentage of Participants With Objective Response as Assessed by the Investigator According to RECIST v1.1 | From randomization until PD, relapse, or death on study from any cause, whichever occurs first (to be assessed according to local standard of care overall up to 5 years)
Duration of Response as Assessed by the Investigator Using RECIST v1.1 | From initial objective response to PD or death on study from any cause, whichever occurs first (to be assessed according to local standard of care overall up to 5 years)
Overall Survival (OS) | From randomization until death from any cause, loss to follow-up, study termination by sponsor, or participant's withdrawal in survival follow-up (overall up to 5 years)
Percentage of Participants With Adverse Events (AE) and Serious Adverse Events (SAEs) | Day 1 Cycle 1 (cycle length=28 days) up to 30 days after last dose of study drug or study discontinuation/termination, whichever is later (overall up to 5 years)
Number of Cycles of Treatment Received for Onartuzumab, Paclitaxel, and Bevacizumab During the Study | Day 1 Cycle 1 (cycle length=28 days) up to last dose of study drug or study discontinuation/termination, whichever is later (overall up to 5 years)
Percentage of Participants With Anti-therapeutic Antibodies (ATAs) Against Onartuzumab | Predose on Day 1 of Cycles 1-4 (cycle length=28 days), 30 days after last administration of onartuzumab or initiation of another therapy (overall up to 5 years)
Serum Levels of ATAs Against Onartuzumab | Predose on Day 1 of Cycles 1-4 (cycle length=28 days), 30 days after last administration of onartuzumab or initiation of another therapy (overall up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (53):
- United States (23):
  - Comprehensive Blood/Cancer Ctr, Bakersfield, California
  - St. Jude Heritage Healthcare; Virgiia K.Crosson Can Ctr, Fullerton, California
  - Can Care Assoc Med Group Inc; Beach Cities Offices, Los Angeles, California
  - Univ of California Los Angeles, Los Angeles, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Sharp Healthcare; Oncology Research Program, San Diego, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists; SCRI, Fort Myers, Florida
  - Suburban Hematology Oncology, Lawrenceville, Georgia
  - Cancer Center of Kansas, Wichita, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute.., Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - North Shore Hem Onc Associates, East Setauket, New York
  - Duke University Medical Center, Durham, North Carolina
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - South Carolina Onc. Associate, Columbia, South Carolina
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - The Sarah Cannon Research Inst, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Northern Utah Associates, Ogden, Utah
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - UZ Antwerpen, Edegem
  - AZ Sint Lucas (Sint Lucas), Ghent
  - CH Jolimont - Lobbes (Jolimont), Haine-Saint-Paul
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - CHU Sart-Tilman, Liège
  - Sint Augustinus Wilrijk, Wilrijk
- France (9):
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Francois Baclesse; Gastro-Enterologie, Caen
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Centre Leon Berard, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut Curie; Oncologie Medicale, Paris
  - Centre Rene Huguenin; CONSULT SPECIALISEES, Saint-Cloud
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
- Germany (4):
  - Praxis Dr. med. Klausmann; SHOD, Aschaffenburg
  - Klinik Johann Wolfgang von Goethe Uni, Frankfurt am Main
  - Klinikum rechts der Isar der TU München; Frauenklinik, München
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
- Spain (5):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona, Barcelona
  - Instituto Catalán de Oncología; Servicio de Farmacia, Barcelona, Barcelona
  - Hospital Universitario Puerta del Mar; Servicio de Oncologia, Cadiz, Cadiz
  - Centro Oncológico Gallego José Antonio Quiroga y Piñeiro, Servicio de Oncologia, A Coruña, La Coruña
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
- United Kingdom (5):
  - Brighton and Sussex Univ Hosp, Brighton
  - Christie Hospital NHS Trust, Manchester
  - The Clatterbridge Cancer Ctr For Oncolgy, Metropolitan Borough of Wirral
  - Mount Vernon Hospital; Centre For Cancer Treatment, Northwood
  - Nottingham City Hospital; Oncology, Nottingham

REFERENCES:
- [Derived] Dieras V, Campone M, Yardley DA, Romieu G, Valero V, Isakoff SJ, Koeppen H, Wilson TR, Xiao Y, Shames DS, Mocci S, Chen M, Schmid P. Randomized, phase II, placebo-controlled trial of onartuzumab and/or bevacizumab in combination with weekly paclitaxel in patients with metastatic triple-negative breast cancer. Ann Oncol. 2015 Sep;26(9):1904-1910. doi: 10.1093/annonc/mdv263. Epub 2015 Jul 22. PMID 26202594